CLINICAL TRIAL: NCT02417441
Title: A Phase IV, Prospective, Randomized, Exploratory, Multicenter, Eeva™ Trial (Time Lapse Eeva - TiLE)
Brief Title: TiLE (Time Lapse Eeva) Clinical Trial
Acronym: TiLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EMR700623_545
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Fertility
Keywords: TiLE; Embryo Assessment; Pregnancy; Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Embryo Viability Assessment + Morphological Grading (Experimental): Embryos of subjects randomized in this group were assessed using Early Embryo Viability Assessment (Eeva) System and morphological grading to identify optimal embryos for transfer.
  Interventions: Device: Eeva
- Morphological Grading (No Intervention): Embryos of subjects randomized in this group were assessed only using morphological grading to identify optimal embryos for transfer.

INTERVENTIONS:
Device: Eeva — Embryos of subjects randomized in this group were assessed using Eeva System and morphological grading to identify optimal embryos for transfer.
  Arms: Early Embryo Viability Assessment + Morphological Grading

SUMMARY:
The purpose of the study was to explore the added value of adjunctive use of Early Embryo Viability Assessment (Eeva) with morphological grading in identifying optimal embryos for transfer.

DETAILED DESCRIPTION:
This study is a Phase IV, open label, prospective, randomized, exploratory, multicenter study. Subjects were randomized in 2:1 ratio to two treatment groups: in the experimental group, embryos were assessed for embryo transfer (ET) with Eeva and morphological grading, while in the control group embryos were assessed with morphological grading only.

ELIGIBILITY:
Inclusion Criteria:

* All infertile subjects treated with In vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI)
* Subject age less than or equal to (<=) 40 years
* Less than or equal to (<=) 3 failed IVF/ICSI cycles
* At least 4 normally fertilized eggs (2 pronuclei [2PN]) in current cycle
* Normal uterine cavity
* Fertilization using only ejaculated sperm (fresh or frozen)
* Subject must have read and signed the Informed Consent Form

Exclusion Criteria:

* Have clinically significant systemic disease
* Have abnormal, undiagnosed gynecological bleeding
* Have any contraindication to Controlled Ovarian Stimulation (COS) for assisted reproductive technologies (ART) and to gonadotropins to be used in ART
* Egg donor cycle
* Planned "freeze all" cycle (oocytes or embryos)
* Concurrent participation in another clinical trial

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 976 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (23):
- Canada (4):
  - Cambrian Wellness Centre, Calgary, Alberta
  - One Fertility, Burlington, Ontario
  - ISIS Regional Fertility Clinic, Mississauga, Ontario
  - Mount Sinai Hospital, Toronto
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - CHRU - Hopital Jeanne de Flandres, Lille
  - Laboratoire Alphabio & Institut de Médecine de la Reproducti, Marseille
  - Hopital Hotel Dieu, Nantes
- Germany (3):
  - Universitatsklinik Schleswig-Holstein, Lübeck
  - Kinderwunsch Centrum München, Munich
  - MVZ Kinderwunschzentrum Wiesbaden GmbH, Wiesbaden
- Italy (4):
  - Montichiari Università degli studi di Bresca, Montichiari
  - Istituto Clinico Humanitas, Rozzano
  - Università degli Studi Torino, Torino
  - Ospedale Versilia, Viareggio
- Telemark hospital Porsgrunn, Skien, Norway
- Spain (3):
  - Clínica Vistahermosa, Alicante
  - Clinica Sagrada Familia, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
- Fertilitetscentrum Stockholm, Stockholm, Sweden
- United Kingdom (3):
  - Bourn Hall, Cambridge
  - Birmingham Women's Health Care NHS Trust, Edgbaston
  - Homerton University Hospital, London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 976 subjects were enrolled, out of which 970 subjects were randomized and started the study.
Period: Overall Study
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading
Started | 645 | 325
Completed | 593 | 306
Not Completed | 52 | 19
Not completed — Inconclusive due to missing data | 52 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading | Total
Number analyzed (Participants) | 645 | 325 | 970
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.6 (3.64) | 33.8 (3.61) | 33.7 (3.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 645 | 325 | 970
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Implantation Rate
Description: Implantation rate was calculated by dividing the number of intrauterine gestational sacs by the number of embryos transferred multiplied by 100.
Time Frame: Gestational Weeks 5 to 8
Population: The intention-to-treat population included all randomized subjects.
Measure: Number (95% Confidence Interval); unit: % of sacs per embryo transferred
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading
Number analyzed (Participants) | 645 | 325
% of sacs per embryo transferred | 30.1 [27.2 to 33.0] | 35.3 [31.1 to 39.5]

2. Secondary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy was confirmed by the presence of a gestational sac with heartbeat as assessed by ultrasonography. Clinical pregnancy rate was measured as the number of clinical pregnancies divided by number of embryo transfer (ET) cycles multiplied by 100.
Time Frame: Gestational Weeks 5 to 8
Population: The intention-to-treat population included all randomized subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of pregnancy per transfer
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading
Number analyzed (Participants) | 645 | 325
Percentage of pregnancy per transfer | 41.0 [37.1 to 44.9] | 47.6 [42.0 to 53.2]

3. Secondary Outcome: Number of Subjects With Ongoing Pregnancy Status
Description: Ongoing pregnancy was defined as having a positive fetal heart beat (FHB) as assessed by ultrasonography at gestational week 10-12. Number of subjects with ongoing pregnancy status has been reported, where "Yes" indicates participants with positive ongoing pregnancy status and "No" indicates participants with negative ongoing pregnancy status .
Time Frame: Gestational Weeks 10 to 12
Population: The intention-to-treat population included all randomized subjects.
Measure: Number; unit: Subjects
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading
Number analyzed (Participants) | 645 | 325
Subjects
  Yes | 30 | 11
  No | 2 | 1
  Missing | 613 | 313

4. Secondary Outcome: Multiple Pregnancy Rate
Description: Multiple pregnancy rate was defined as a clinical pregnancy with greater than equals to (>=) 2 fetal sacs as assessed by ultrasonography. Multiple Pregnancies rate was measured by number of multiple pregnancies divided by number of embryo transfer cycles multiplied by 100.
Time Frame: Gestational Weeks 5 to 8
Population: The intention-to-treat population included all randomized subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of pregnancy per transfer
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading
Number analyzed (Participants) | 645 | 325
Percentage of pregnancy per transfer | 6.4 [4.5 to 8.3] | 8.4 [5.3 to 11.5]

5. Secondary Outcome: Utilization Rate
Description: Utilization rate was defined as the sum of number of transferred and frozen embryos divided by number of normally fertilized oocytes multiplied by 100.
Time Frame: Day 3 or Day 5/6 of embryo culture
Population: The intention-to-treat population included all randomized subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of embryos
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading
Number analyzed (Participants) | 645 | 325
Percentage of embryos | 48.6 [47.1 to 50.1] | 49.6 [47.5 to 51.7]

6. Secondary Outcome: Spontaneous Miscarriage Rate
Description: Spontaneous miscarriage rate was measured by the number of spontaneous miscarriages as communicated during medical appointment or by telephone contact divided by number of clinical pregnancies multiplied by 100.
Time Frame: Gestational Weeks 10 to 12
Population: The intention-to-treat population included all randomized subjects.
Measure: Number; unit: Percentage of miscarriages
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading
Number analyzed (Participants) | 645 | 325
Percentage of miscarriages | NA — Technical issues of eCRF led to incorrect and misleading data which was excluded and hence, no accurate data is available for this outcome measure. | NA — Technical issues of eCRF led to incorrect and misleading data which was excluded and hence, no accurate data is available for this outcome measure.

7. Other Pre Specified Outcome: Eeva Conformity in Early Embryo Viability Assessment + Morphological Grading Group for Day 3 Embryo Transfer (ET)
Description: Eeva Conformity was reported as the number of subjects who were compliant to use Eeva in embryo assessment in the "Early Embryo Viability Assessment + morphological grading" group. Eeva-compliance subgroup refers to subjects whose embryos were assessed by embryologists following the recommendation of Eeva system and the instructions for use (IFU) of Eeva. Subgroup analysis revealed a high incidence of Eeva noncompliance in the experimental group, which compromised the quality of this study. Only "Early Embryo Viability Assessment + Morphological Grading" reporting arm was applicable for this outcome measure.
Time Frame: Day 3 of embryo culture
Population: Subgroup Analysis Set included subjects from "Early Embryo Viability Assessment + morphology grading" group for whom the embryologist has followed the recommendation of the Eeva system. Here, Number of Subjects analyzed signifies those who were evaluable for this outcome measure.
Measure: Number; unit: Subjects
Arm/Group | Early Embryo Viability Assessment + Morphological Grading
Number analyzed (Participants) | 242
Subjects | 163

8. Other Pre Specified Outcome: Eeva Conformity in Early Embryo Viability Assessment + Morphological Grading Group for Day 5/6 Embryo Transfer (ET)
Description: Eeva Conformity was reported as the number of subjects who were compliant to use Eeva in embryo assessment in the "Early Embryo Viability Assessment + morphological grading" group. Eeva-compliance subgroup refers to subjects whose embryos were assessed by embryologists following the recommendation of Eeva system and the IFU of Eeva. Subgroup analysis revealed a high incidence of Eeva noncompliance in the experimental group, which compromised the quality of this study. Only "Early Embryo Viability Assessment + Morphological Grading" reporting arm was applicable for this outcome measure.
Time Frame: Day 5/6 of embryo culture
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Early Embryo Viability Assessment + Morphological Grading
Number analyzed (Participants) | 191
Subjects | 87

9. Post Hoc Outcome: Number of Sites With Subjects Reporting Fetal Heart Beat (FHB) Positive Implantation Rate (IR)
Description: Number of sites with subjects reporting fetal heart beat (FHB) positive implantation rate (IR) were reported. Overall combined data for "Early Embryo Viability Assessment + Morphological Grading" and "Morphological Grading" arm was planned to be reported.
Time Frame: Gestational Weeks 5 to 8
Population: Subgroup analysis set included subjects reporting positive fetal heart beat implantation rate from both "Early Embryo Viability Assessment and Morphological grading arm" and "Morphological grading arm". Here, Number of Subjects analyzed signifies those who were evaluable for this outcome measure.
Measure: Number; unit: Sites
Units Other Than Participants: Sites
Groups:
- All Subjects (FHB Positive IR): All subjects with positive fetal heart beat (FHB) implantation rate (IR) from "Early Embryo Viability Assessment + Morphological Grading" and "Morphological Grading" arm were randomized in this group.
Arm/Group | All Subjects (FHB Positive IR)
Number analyzed (Participants) | 649
Number analyzed (Sites) | 15
Sites
  Day 3 of embryo transfer: number analyzed (Participants) | 359
  Day 3 of embryo transfer: number analyzed (Sites) | 12
  Day 3 of embryo transfer | 5
  Day 5/6 of embryo transfer: number analyzed (Participants) | 290
  Day 5/6 of embryo transfer: number analyzed (Sites) | 14
  Day 5/6 of embryo transfer | 7

ADVERSE EVENTS:
Time Frame: Not Applicable (NA)
Description: This is a fertility device technology study and this study was not designed to monitor all-cause mortality, serious, and other (not Including serious) adverse events. Therefore, all-cause mortality, serious, and other (not Including serious) adverse events data could not be reported.
Arm/Group | Early Embryo Viability Assessment + Morphological Grading | Morphological Grading
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Subgroup analysis revealed high incidence of Eeva noncompliance in the experimental arm and heterogeneous results across sites. Thus, no decisive conclusion can be made from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT02417441/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT02417441/SAP_001.pdf